CLINICAL TRIAL: NCT07163871
Title: The Effect of Individualized Home Visits Under the Supervision of Midwives on Maternal Functioning, Breastfeeding, and Resilience: a Randomized Controlled Trial
Brief Title: Breastfeeding, Maternal Functioning, and Resilience
Acronym: MLIHV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medine Yönder (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Sponsor-Investigator, Medine Yönder, MSc Student, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Hatice Gül ÖZTAŞ
Record Dates: First submitted 2025-08-19; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Women
Keywords: breastfeeding; midwifery; postpartum depression; home visit
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum | interventions — Milk, Human

STUDY DESIGN:
Intervention Model Description: One group received training, while the other group was surveyed without receiving training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): This group was given detailed information on postpartum hygiene, breastfeeding, baby care, breast milk, and other necessary topics.
  Interventions: Behavioral: Postpartum hygiene, breast milk, and breastfeeding education have been provided for new mothers.
- control group (No Intervention): No training other than routine postnatal training has been provided. No intervention has been made.

INTERVENTIONS:
Behavioral: Postpartum hygiene, breast milk, and breastfeeding education have been provided for new mothers. — During the first ten days after birth, the first month, and the third month, new mothers received detailed care and education through home visits in addition to routine postnatal education. Information was shared at the mother's request as needed.
  Arms: intervention group

SUMMARY:
This study aims to examine the effect of individualized home visits led by midwives on maternal functioning, breastfeeding attitudes, and depression levels.

DETAILED DESCRIPTION:
Childbirth is one of the most unique and important events in a woman's life. The postpartum period is defined as the period that begins immediately after childbirth and ends six weeks later. The period corresponding to the first twenty-four hours is called the immediate period; the period from the first twenty-four hours to the end of the first week is called the early period; and the period from the second week after childbirth to the end of the sixth week is called the late period. We can say that the postpartum period is a critical period for women, newborns, and other family members. For primiparous women, it is a very challenging process that requires adaptation to new roles and brings with it emotional, physical, social, and spiritual changes and confusion.

The postpartum period is also a transition period during which women and family members must adapt to new physical, psychological, and social circumstances In many developed countries, the hospital stay after vaginal delivery is typically less than 48 hours during this transition period. In Turkey, the hospital stay for the mother and newborn is a maximum of 24 hours after a normal birth and 48 hours after a cesarean section . However, this period is quite short in terms of providing education related to the postpartum period, monitoring potential complications, and addressing psychological issues. In this context, home visits are of great importance for the early detection and intervention of difficulties faced by women who cannot access adequate healthcare services, for educating them on how to care for themselves and their babies, and for providing other personal care services. Home visits during the postpartum period contribute to the protection and improvement of the mother's health by providing technical, psychological, and therapeutic support regarding her care, education, and needs at home.

The World Health Organization (WHO) recommends at least four follow-up visits for all mothers and newborns within six weeks after birth. These should be conducted on the 1st day (first 24 hours), 3rd day (48-72 hours), 7-14th days, and 30-42nd days . It is believed that face-to-face physical examinations and/or screenings of the mother and newborn are more effective during these follow-ups. Midwives can provide personalized postpartum care through home visits tailored to the needs of the mother and newborn. Midwife-led postpartum care is an important public health intervention for women, newborns, and other family members . Midwife-led postpartum home visits can increase awareness among mothers regarding breastfeeding initiation, breastfeeding continuation, manual milk expression and proper milk storage, family planning and postpartum contraception, lochia monitoring, home hygiene, and newborn care .

Unfortunately, there is currently no strong evidence that home visits improve postpartum maternal and infant health, and there is a need for evidence-based research on these topics . Research on midwife-led postpartum home visits and home care is not at the desired level. A Swedish study examining the postpartum care experiences of first-time mothers after discharge from the hospital showed that midwives played a supportive role and increased parents' self-confidence . A Norwegian study on women's experiences of home visits by midwives in the early postpartum period identified three main themes: relational continuity, postpartum conversation, and vulnerability . A study conducted in the UK found that pregnancy, childbirth, and postpartum care were associated with improved health outcomes for women and babies in socially disadvantaged and diverse communities. A home visitation program conducted in Australia for vulnerable families in disadvantaged areas demonstrated improvements in participants' parenting skills and well-being, participation in community networks, and access to support services . In Sweden, vulnerable women who received long-term home visits reported improved parenting skills and increased confidence when discussing issues with professionals . A longitudinal study investigating the impact of home visits in Germany also reported improvements in the skills of mothers receiving care in areas such as newborn care, managing family relationships, and seeking, receiving, and accepting external help .

Becoming a mother is a physiological process in which behaviors specific to women and different from the norm are observed. The transition to motherhood can be considered an important developmental event in a woman's life . The process of assuming the role of motherhood should begin during pregnancy and continue until the birth of the baby . Although the role of motherhood begins during pregnancy, it truly begins after the baby is born, when the mother becomes aware of her maternal functions, roles, and responsibilities through interaction with the baby . The success of the maternal role indicates the quality of parenting behaviors and has a significant impact on the social development of the newborn. The formation of maternal identity also contributes to a woman's psychosocial development .

Breastfeeding is one of the actions that not only affects the growth and development of the baby but also the health of the family and society . Breastfeeding provides babies with the nutrients they need for healthy growth and development in the best possible way. The World Health Organization (WHO) recommends that mothers exclusively breastfeed their children for the first six months of life and continue breastfeeding with complementary foods until the age of two or beyond. However, approximately 40% of infants worldwide are exclusively breastfed during the first six months of life . At the national level in Turkey, this rate is similar. Breastfeeding rates among women are influenced by many factors, including sociodemographic characteristics, psychosocial factors, attitudes toward breastfeeding, knowledge about breastfeeding, and self-efficacy in breastfeeding .

Women may experience some psychological distress due to the effects of postpartum hormones. The most common psychological disorder during this period is postpartum depression. Postpartum depression is defined as a mood disorder that can last from the first 2-4 weeks after birth to the first year . Although it cannot be attributed to a single cause, it is thought to be caused by genetic predisposition, hormonal imbalances, and psychological and physiological factors during this process . The symptoms of postpartum depression vary from mother to mother, but they can include sleep problems, inability to enjoy life, unexplained weight loss, feelings of inadequacy, guilt, tension, and thoughts of suicide . When considering the causes of postpartum depression, unexpected health problems, insufficient social support, health problems in the newborn, a history of psychiatric illness, the type of delivery, the number of births, and, in addition, the woman's birth experience, how she perceives the birth, and how she records it in her memory are among the influencing factors.

Similar studies have been conducted in the literature. Bostancı Daştan and colleagues examined the mental health of pregnant women through home visits and emphasized that pregnancy can cause crisis and that depression symptoms should be detected as early as possible. Erenel and Eroğlu conducted an experimental study to determine the effect of a breastfeeding education model supported by home visits in the early postpartum period on effective breastfeeding behavior. They found that a large proportion of the women participating in the study continued effective breastfeeding, while the rate of effective breastfeeding in the control group was much lower. In the experimental study conducted by Demir Yıldırım and Hotun Şahin, it was determined that home visits during pregnancy monitoring were an effective model in increasing pregnant women's knowledge about the prenatal period, their desire for vaginal delivery, and the duration of initial and subsequent breastfeeding. However, no study has been found in the literature regarding the effect of individualized home visits on maternal function, breastfeeding attitudes, and depression levels. The aim of this planned study is to support the postpartum care process conducted at the primary care level through home visits led by midwives and to observe its effect through a control group. The home visits are intended to increase satisfaction with the services provided during the postpartum period, ensure the provision of quality postpartum care, and thereby minimize the risk of bleeding and infection and facilitate adaptation to motherhood. In addition, the aim is for women to receive the necessary education about the postpartum period, to perform postpartum self-care appropriately, to meet the feeding and care needs of the newborn, to increase their self-efficacy in breastfeeding, and to minimize the risk of postpartum depression.

ELIGIBILITY:
* 18 yaş ve üzerinde,
* Primipar,
* Miadında doğum yapmış,
* Sağlıklı tek bebek dünyaya getiren,
* Psikiyatrik bir tanı almamış olan,

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is being conducted on women who have recently given birth.
Enrollment: 94 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Barkin Maternal Function Scale | 2 week
  It was developed by Barkin in 2009 to assess functional status during the postpartum period. The validity and reliability study of the Turkish version of the scale was conducted by Aydın and Kukulu (2016) (Aydın, Kukulu, 2016). The scale consists of 16 items divided into five subscales: self-care (3 items), maternal psychology (2 items), infant care (4 items), social support (3 items), and adjustment to motherhood (4 items). The items on the scale are 7-point Likert-type and numbered from 0 to 6. The responses are as follows: 0 "I completely disagree," 1 "I disagree," 2 "I somewhat disagree," 3 "I am undecided," 4 "I somewhat agree," 5 "I agree," and 6 "I completely agree." The lowest possible score on the scale is 0, and the highest possible score is 96 (Aydın & Kukulu, 2018). A high score on the scale indicates that the individual has a high level of maternal functioning. In Aydın and Kukulu's study, the Cronbach's alpha reliability coefficient of the scale was found to be 0.73.

SECONDARY OUTCOMES:
LATCH Breastfeeding Assessment Scale | 2 week
  LATCH breastfeeding assessment and evaluation scale Evaluation Criterion Meaning of Evaluation Criterion L Latch on Breast Baby latching onto the breast A Audible Swallowing Visible swallowing movements of the baby T Type of Nipple Type of nipple C Comfort of Breast/Nipple Mother's comfort with her breast/nipple H Hold/Position Mother's position when holding the baby Each criterion that makes up LATCH is scored on a scale of 0, 1, or 2, with a total possible score of 10. There is no cutoff point for the scale. Breastfeeding is evaluated by summing the scores. A low score on the scale indicates a need for support and monitoring regarding breastfeeding. As the scale score increases, it is understood that breastfeeding success is high (Appendix 4). The Cronbach's alpha value of the scale was found to be 0.95 by Yenal and Okumuş (2003), 0.94 by Demirhan (1997), and 0.96 by Koyun (2001) (Demirhan, 1997; Koyun, 2001; Yenal and Okumuş, 2003).
Infant Feeding Attitude Scale | 2 week
  The Infant Feeding Attitude Scale was developed to assess women's attitudes toward breastfeeding and to estimate the duration of breastfeeding as well as the choice of infant feeding method (de la Mora et al. 1999). The scale consists of 17 items on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Nine items on the scale relate to breast milk, and eight items relate to formula milk. Formula milk items are reverse-scored (1=5, 2=4, 4=2, and 5=1). The total attitude score ranges from 17 to 85 points. The Cronbach's alpha coefficient of the scale was found to be 0.86 (de la Mora et al., 1999). The validity and reliability of the scale in Turkish were established by Ekşioğlu and colleagues (2016). The Cronbach's alpha internal consistency coefficient of the scale was determined to be 0.71 (Ekşioğlu et al., 2016). In this study, the Cronbach's alpha internal consistency coefficient of the scale was calculated as 0.72.
Edinburgh Postpartum Depression Scale | 2 week
  The validity and reliability of the scale in Turkish were established by Engindeniz, and the Cronbach's alpha value of the scale was determined to be 0.79 (Engindeniz, 1996). The scale is used to determine the risk of depression in the postpartum period and to measure changes in its level and severity. The EPDÖ is a self-assessment scale consisting of 10 items that reflect the individual's psychological state over the past seven days. Each item is scored on a 0-3 scale with a four-point Likert scale: "Yes, always," "Yes, most of the time," "No, not very often," and "No, never." The lowest possible score on the scale is 0, and the highest possible score is 30. Items 1, 2, and 4 are scored as 0, 1, 2, 3, while items 3, 5, 6, 7, 8, 9, and 10 are scored in reverse as 3, 2, 1, 0. The cutoff point for the EPDÖ is calculated as 12/13, and the total score indicates the severity of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü Imam Univercity, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF